CLINICAL TRIAL: NCT02722148
Title: Application of a Novel Allergen-Specific Immune Signature Directed Approach to Dietary Elimination Therapy in Patients With Eosinophilic Esophagitis (IDiET)
Acronym: IDiET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-2719
Record Dates: First submitted 2016-03-24; First posted 2016-03-29 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2018-08

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; Diet Elimination Therapy
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Enrolled Patients (Experimental): All enrolled subjects will receive a novel allergen-specific immune signature directed approach to dietary elimination therapy
  Interventions: Device: Novel Allergen-Specific Immune Signature Directed Approach to Dietary Elimination Therapy

INTERVENTIONS:
Device: Novel Allergen-Specific Immune Signature Directed Approach to Dietary Elimination Therapy — A novel assay developed by the investigator to diagnose food allergens. Results from the assay are used to guide food elimination therapy for the treatment of Eosinophilic Esophagitis (EoE).

SUMMARY:
This is a prospective single center clinical trial of allergen-specific immune signature-guided dietary elimination therapy to assess the clinical effectiveness of this technique.

DETAILED DESCRIPTION:
This is a prospective single center clinical trial of allergen-specific immune signature-guided dietary elimination therapy to assess the clinical effectiveness of this technique.

Potential subjects will be approached regarding the study. If eligible and interested, then informed consent will be obtained and they will be enrolled in the study. If the subject as had an esophagogastroduodenoscopy (EGD) at UNC with 3 month since enrollment, clinical biopsies from the EGD show active EoE and the subject continues to meet consensus guidelines for active EoE, and research biopsies were taken during that EGD that can be used for this study, then the subject will complete questionnaires and a blood draw only. The blood draw may be abbreviated if the subject had research blood drawn during the same recent EGD that can be used in this study.

If subjects have not had an EGD with biopsies at UNC within 3 months prior to enrollment, then they will complete questionnaires, a blood draw, and be scheduled to receive a routine care esophagogastroduodenoscopy (EGD) at UNC facilities with clinical and research biopsies. However, in some cases, samples that were obtained prior to this time frame can be used, as long as the samples were obtained when the EoE was active and there were no major changes in clinical status.

During the routine care endoscopy, clinical biopsies will be taken for routine care purposes, and additional research biopsies will be collected for research purposes for diet elimination testing and to be stored for future research studies from the distal, mid, and proximal esophagus. Blood will also be collected during this visit, and questionnaires completed. If research biopsies are unable to be obtained during this EGD the subject will no longer continue in the study and will be considered a screen fail. If pathology from routine care biopsies does not confirm a diagnosis of active EoE, then the subject will no longer continue in the study and will be considered a screen fail. If subjects have had an EGD with clinical and research biopsies within 3 months prior to enrollment, then research biopsies taken during that EGD will be used for this study. As noted above, in some cases, samples that were obtained prior to this time frame can be used, as long as the samples were obtained when the EoE was active and there were no major changes in clinical status.

After completion of the EGD (or collection of EGD records and previous biopsies if an EGD was previously completed), and confirmation of eligibility, subjects will be scheduled for a routine care nutrition counseling appointment. Two weeks prior to the routine care nutrition counseling appointment, subject will begin the dysphagia symptom questionnaire (DSQ). During the routine care nutrition counseling appointment, the subject will receive counseling on which foods to eliminate based on the novel assay results from the research biopsies. Subjects will also receive an allergy skin test during this visit. Results from the allergy skin test will not be used to drive food elimination diet.

Subjects will follow their assigned food elimination diet for 6 weeks. At 6 weeks subjects will be scheduled for a routine care esophagogastroduodenoscopy (EGD) with biopsies for clinical purposes. Two weeks prior to the 6 week EGD subjects will restart the DSQ. Data will be collected from the 6 week EGD but no research specific biopsies will be obtained during that visit. Research specific blood will be taken at this visit. Study participation is complete after completion of the 6 week EGD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-80 years old
2. Meet one of the following:

   1. Active EoE as per consensus guidelines OR
   2. Undergoing upper endoscopy for a clinical suspicion of EoE
3. No prior history of dietary elimination therapy

Exclusion Criteria:

1. Concomitant eosinophilic gastroenteritis
2. Any corticosteroid exposure in the 4 weeks prior to their baseline endoscopic exam
3. Previous esophageal surgery
4. Medical instability that precludes safely performing upper endoscopy
5. Inability to read or understand English
6. Pregnant women

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan S Dellon, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share data

REFERENCES:
- [Derived] Dellon ES, Guo R, McGee SJ, Hamilton DK, Nicolai E, Covington J, Moist SE, Arrington A, Wright BL, Burks AW, Vickery BP, Kulis M. A Novel Allergen-Specific Immune Signature-Directed Approach to Dietary Elimination in Eosinophilic Esophagitis. Clin Transl Gastroenterol. 2019 Dec;10(12):e00099. doi: 10.14309/ctg.0000000000000099. PMID 31789931

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enrolled Patients
Started | 24
Completed | 19
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Non compliant with treatment regimen | 3

BASELINE CHARACTERISTICS:
Population: Data unavailable for two participants who were lost to follow-up.
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Histologic Responders
Description: The primary outcome will be histologic response, defined as a post-treatment esophageal eosinophil count of <15 eos/hpf.
Time Frame: 6 Weeks
Population: Data reported only for compliant participants
Measure: Number; unit: percentage of participants
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 19
percentage of participants | 21

2. Secondary Outcome: Median Peak Esophageal Eosinophil Count
Description: Eosinophil count per High Power Field
Time Frame: 6 Weeks
Measure: Median (Inter-Quartile Range); unit: eosinophils per high power field
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 19
eosinophils per high power field | 35 [20 to 63]

3. Secondary Outcome: Endoscopy Score
Description: Post treatment endoscopic appearance, as measured by a validated endoscopy score - the EoE Endoscopic Reference Score (EREFS). This score measures endoscopic severity with a set of five endoscopic findings (exudates, rings, edema, furrows, and strictures), and ranges from 0-9, with higher scores indicating higher endoscopic severity.
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 19
units on a scale | 3.0 (1.9)

4. Secondary Outcome: Dysphagia Symptom Score
Description: Post treatment symptoms, as measured by a validated dysphagia symptom score, the EoE Symptom Activity Index (EEsAI). This score ranges from 0-100, with higher scores indicating more severe symptoms. A score of < 20 indicates clinical remission.
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 19
score on a scale | 25.0 (23.1)

ADVERSE EVENTS:
Time Frame: Baseline through post treatment assessments (approximate total of 6 weeks).
Arm/Group | Enrolled Patients
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT02722148/Prot_SAP_000.pdf